CLINICAL TRIAL: NCT01016678
Title: Early Intervention, Randomized, Mulitcenter, Placebo-Controlled, 4-Period Crossover, Multi-Attack Study to Evaluate Efficacy & Safety of ComboProduct Containing Sumatriptan and Naproxen Sodium for Acute Treatment of Migraine in Adolescents
Brief Title: Treximet Early Intervention Adolescent Migraine
Acronym: TEAM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Premiere Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TEAM2009
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — sumatriptan-naproxen; Sumatriptan; Naproxen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Active, Active, Active, Placebo (Other): One fifth of the 105 subjects will be randomized to this arm and treat their four migraines in this order. First three will be treated with Active Treximet and the last or 4th migraine will be treated with Placebo.
  Interventions: Drug: Treximet; Drug: Placebo
- Active, Active, Placebo, Active (Other): This is another of the five treatment arms. One fifth of the 105 subjects will be randomized to this group and will treat the first two migraines with Active drug, Treximet, and then the third migraine with placebo and the last (4th) migraine with Treximet.
  Interventions: Drug: Treximet; Drug: Placebo
- Active, Placebo, Active, Active (Other): Approximately one fifth of the 105 subjects will be randomized to this group and treat their first migraine with Active Treximet and the second migraines with Placebo. The final two migraines treated will be with Active study drug.
  Interventions: Drug: Treximet; Drug: Placebo
- Placebo, Active, Active, Active (Other): One fifth of the 105 subjects will be randomized to this treatment arm, where they will treat the first headache with placebo and the remaining three migraines will be treated with Active treximet.
  Interventions: Drug: Treximet; Drug: Placebo
- Active, Active, Active, Active (Other): One fifth of the subject will treat all their migraines with Active Treximet.
  Interventions: Drug: Treximet

INTERVENTIONS:
Drug: Treximet — 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
  Other Names: Imitrex and Naproxen Sodium
Drug: Placebo — Dummy pill comparator
  Other Names: Sugar Pill
  Arms: Active, Active, Active, Placebo; Active, Active, Placebo, Active; Active, Placebo, Active, Active; Placebo, Active, Active, Active

SUMMARY:
The study involves approximately 105 adolescent (ages 12-17) subjects to be screened at 4 sites across the US. All subjects enrolled will treat up to 4 MILD migraines over a 6 month period. They will be required to have three office visits during the six months. All subjects will be randomized to either Treximet (85mg Imitrex/500mg Naproxen Sodium) or Placebo (sugar-pill) in four of the five treatment arms with a 3 to 1 ratio. A fifth treatment arm will treat all 4 migraines with active drug, Treximet. The hypothesis is that Treximet will prove to be a safe and effective treatment for this population, that has so few treatment for migraine. And Treximet will be superior over placebo for pain free endpoints at 2 and 24 hours.

DETAILED DESCRIPTION:
There are two primary treatment comparisons for this study: 1) the percentage of subjects' pain free at 2 hours after treatment with TREXIMET versus placebo across attacks, and 2) the percentage of subjects who are sustained pain free at 24 hours after treatment with TREXIMET versus placebo across attacks.

The following alternative hypothesis will be tested to see if there is a difference in the proportion of subjects who are pain free at 2 hours with TREXIMET versus placebo at all attacks, OR there is a difference in the proportion of subjects who are sustained pain free at 24 hours with TREXIMET versus placebo at all attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 12-17.
2. Subject has migraine with or without aura (ICHD-II criteria, 1.2.1 or 1.1). A history of at least 1 but no more than 8 attacks per month on average over the past 6 months prior to screening visit. Attacks should be moderate to severe and last for at least 3 hours.
3. Subject is able to distinguish migraine from other headaches and can determine when a mild headache will become a moderate/severe migraine.
4. Female subjects are eligible for participation provided they are of non-child bearing potential or if started menses; they are on a stable regimen of approved contraception.
5. Subject and subject's parent or legal guardian are able to read and write English.
6. Subject is able to read, comprehend, and complete subject diaries.
7. Subjects' parent or legal guardian is willing and able to provide Informed Consent prior to subject entry into the study.
8. Subject is willing and able to provide Informed Assent prior to entry into the study.

Exclusion Criteria

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Subject is < 74 pounds (33.3kg) and no greater than 260lbs (117.9kg)
2. Subject has greater than or equal to 15 headache days per month in total.
3. Subject has secondary headaches i.e. complex migraine, hemiplegic, or basilar.
4. Subject, in investigators opinion is likely to have unrecognized cardiovascular or cerebrovascular disease.
5. Subject has uncontrolled hypertension at screening or is taking an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker.
6. Subject has a history of congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in the study.
7. Subject has evidence or history of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease, or signs/symptoms consistent with the above.
8. Subject has a evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold, or has been treated with an anti-epileptic drug for seizure control within 5 years prior to screening.
9. Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study.
10. Subject has a hypersensitivity, allergy, intolerance, or contraindication to the use any triptan, NSAID, or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps or asthma.
11. Subject has used an ergot medication in the previous three months for migraine prophylaxis or is taking a medication that is not stabilized for at least two months for either chronic or intermittent migraine prophylaxis or other co-morbid condition.
12. Subject has taken or plans to take a monoamine oxidase inhibitor (MAOI) including herbal preparations containing St. Johns Wort (Hypericum perforatum), anytime within the two weeks prior to screening and two weeks past exit of study.
13. Subject has a history of any bleeding disorder or is currently taking any anti-coagulant or any antiplatelet agent.
14. Subject has evidence or history of any gastrointestinal surgery, GI ulceration, or perforation in the past six months, gastrointestinal bleeding in the past year, or evidence or history of inflammatory bowel disease.
15. Subject is pregnant, actively trying to become pregnant, or breast feeding or Subject is not willing to have pregnancy test(s).
16. Subject has evidence of illicit drug or alcohol abuse within the last year or any concurrent psychiatric condition which, in the investigator's opinion, will likely interfere with study conduct and participation in the trial.
17. Subject has participated in any investigational drug trial within the previous 4 weeks or plans to participate in another study at any time during this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul K Winner, DO, Principal Investigator — Premiere Research Institute; Andrew Hershey, MD, Principal Investigator — Cincinnati Childrens Hospital; Steve L Linder, MD, Principal Investigator — Dallas Pediatric Neurology Associates; Donald W Lewis, MD, Principal Investigator — Children's Hospital of The King's Daughters
Locations (4):
- United States (4):
  - Premiere Research Institute, West Palm Beach, Florida
  - Andrew Hershey, Cincinnati, Ohio
  - Steve L. Linder, Dallas, Texas
  - Don W. Lewis, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
There is no plan in place to enter every single patient in separtely

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment period started in March 2010 and the last subject was exited March 2013. The 4 sites who recruited all patients, consisted of 2 private practices and 2 children's hospital based site.
Pre-assignment Details: 104 patients were randomized and dispensed study drug but only 94 of those patients actually treated at least one migraine, so therefore 94 subjects data was used in the analysis.
Groups:
- Active, Active, Active, Placebo: Treximet: 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
  First three migraines will be treated with Active Treximet and the last 4th migraine will be treated with Placebo
- Active, Active, Placebo, Active: Treximet: 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
  First two migraines will be treated with Active Treximet and then the 3rd migraine will be treated with Placebo and the last 4th migraine will be treated with Treximet
- Active, Placebo, Active, Active: Treximet: 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
  The first migraine will be treated with Active Treximent and the second migraine with Placebo. The final two migraines will be treated with Active Treximet
- Placebo, Active, Active, Active: Treximet: 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
  First migraine will be treated with Placebo and the last three migraines will be treated with Active Treximet
- Active, Active, Active, Active: Treximet: 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
  All migraines (up to four) will be treated with active treximet
Period: Overall Study
Arm/Group | Active, Active, Active, Placebo | Active, Active, Placebo, Active | Active, Placebo, Active, Active | Placebo, Active, Active, Active | Active, Active, Active, Active
Started | 20 | 17 | 19 | 19 | 19
Completed | 18 | 14 | 15 | 19 | 13
Not Completed | 2 | 3 | 4 | 0 | 6

BASELINE CHARACTERISTICS:
Population: 104 subjects were randomized in the study but only 94 subjects actually dosed with study drug and completed at least one diary assessment post dose.
Groups:
- Adolescents Age 12-17: All subjects were adolescent males and females with diagnosis of Migraine and a frequency of 1-8 migraines per month on average
Arm/Group | Adolescents Age 12-17
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 104
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.8 [12 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 2-hour Pain Free Active Study Drug
Description: All data was collected and measured from self-reported patient diaries
Time Frame: 3 years
Population: The number of subjects randomized to treatment was 104, which included 94 subjects who treated at least one migraine with study drug and were included in the safety and efficacy data analysis
Measure: Number; unit: Participants
Groups:
- Migraine Attack 1; Migraine Attack 2; Migraine Attack 3; Migraine Attack 4: The participants were instructed to treat 4 migraine attacks in the trial and according to the randomization schedule could potentially treat 3 attacks with active study drug (sumatriptan/naproxen sodium) and 1 attack with placebo, with different placement of the placebo for every 10 subjects. There are also a group of subjects in which all attacks were treated with active study drug.
  Treximet: 85mg Imitrex with 500mg Naproxen Sodium combination tablet for treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hours period.
Arm/Group | Migraine Attack 1 | Migraine Attack 2 | Migraine Attack 3 | Migraine Attack 4
Number analyzed (Participants) | 94 | 90 | 82 | 81
Participants
  Pain Free at 2 hours post dose for Active Treatmen | 35 | 23 | 21 | 24
  Pain Free at 2 Hours Post Dose for Placebo | 2 | 2 | 3 | 6
Statistical Analysis 1: Comparison: Migraine Attack 1 vs Migraine Attack 2 vs Migraine Attack 3 vs Migraine Attack 4; Comparison of percentage of participants pain free at 2 hours post-dose (active) to percentage of participants pain free at 2 hours post-dose (placebo); Test type: Superiority or Other; p = 0.0038, Chi-squared; Difference in percentages = 18

2. Primary Outcome: Percentage of Migraine Attacks With Sustained Pain Free Response From 2 to 24 Hours Post-Dose
Description: All data was collected and measured from self-reported patient diaries
Time Frame: 3 years
Population: Patients who treated with study drug and were pain free at 2 hours and then continued to be pain free through 24 hours
Measure: Number; unit: percentage of attacks
Units Other Than Participants: Migraines
Groups:
- Active Drug: Treximet 85mg Imitrex with 500mg Naproxen Sodium combination tablet for the treatment of migraine headache. The adult dosage is 1 tab Q12H for migraine and no more than 2 tablets in a 24 hour period.
- Placebo: Equivalent looking pill just like Treximet but only containing sugar, "sugar pill".
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 54 | 13
Number analyzed (Migraines) | 103 | 13
percentage of attacks | 86 | 78
Statistical Analysis 1: Comparison: Active Drug vs Placebo; Test type: Superiority or Other; p = 0.1294, Chi-squared; difference in percentages = 8

3. Primary Outcome: Percentage of Migraine Attacks With Pain Free Response at 2 Hours Post-Dose Following Early Intervention
Description: All data was collected and measured from self-reported patient diaries
Time Frame: 3 years
Population: 94 subjects treated at least one migraine attack with active drug or placebo were analyzed while only 74 subjects had the potential to take placebo during one of their 4 migraine attacks
Measure: Number; unit: percentage of attacks
Units Other Than Participants: number of migraine attacks
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 94 | 74
Number analyzed (number of migraine attacks) | 277 | 70
percentage of attacks | 32 | 18

4. Secondary Outcome: To Evaluate the Consistency of Response Across Four Migraine Attacks at 1, 2, 4, and 24 Hours After Treatment. Frequency of Rescue Medications Needed and the Consistency of Other Symptom Relief i.e. Nausea, Vomiting, Photophobia, and Phonophobia.
Description: Collected from patient reported paper diaries
Time Frame: 3 years
Population: This analysis data was not collected.
Arm/Group | Active, Active, Active, Placebo | Active, Active, Placebo, Active | Active, Placebo, Active, Active | Placebo, Active, Active, Active | Active, Active, Active, Active
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Entire Study 3 years
Description: All adverse events are reported here whether patient had taken active drug or placebo and it is not separated per intervention
Arm/Group | Active, Active, Active, Placebo | Active, Active, Placebo, Active | Active, Placebo, Active, Active | Placebo, Active, Active, Active | Active, Active, Active, Active
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/17 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 2/20 | 8/17 | 5/19 | 8/19 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active, Active, Active, Placebo (N=20) | Active, Active, Placebo, Active (N=17) | Active, Placebo, Active, Active (N=19) | Placebo, Active, Active, Active (N=19) | Active, Active, Active, Active (N=19)
Prolonged Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient was treated in the hospital for a prolonged migraine but it was not related to study drug. Study drug was taken 10 days prior to event onset.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active, Active, Active, Placebo (N=20) | Active, Active, Placebo, Active (N=17) | Active, Placebo, Active, Active (N=19) | Placebo, Active, Active, Active (N=19) | Active, Active, Active, Active (N=19)
Neck Spasm/Tension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 2 (4) — The percentage of occurrence was 6.4%
Drowsiness (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (3) — The percentage of occurrence was 4.3%
Throat tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (6) — The percentage of occurrence was 5%
Stiff Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) — Tightness or Stiff feeling in jaw
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Tongue Swelling (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) — Numbness in Extremities
Burning Sensation Face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Poison Ivy Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bad Taste (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Simplex Right Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abcess Right Leg (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bruised Coccyx (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Broken Right Arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weird Feeling, Out of Body Sensation (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No